CLINICAL TRIAL: NCT00000538
Title: Dietary Effects on Lipoproteins and Thrombogenic Activity
Acronym: DELTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 81; U01HL049644 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2014-08

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Coronary Heart Disease Risk Reduction; Heart Diseases; Hyperlipoproteinemia; Myocardial Ischemia; Thrombosis
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Diseases; Hyperlipoproteinemias; Myocardial Ischemia; Thrombosis | interventions — Diet, Fat-Restricted

INTERVENTIONS:
Behavioral: diet, fat-restricted

SUMMARY:
To evaluate the effects of carefully controlled diets on lipoproteins and clotting factors in different demographic groups.

DETAILED DESCRIPTION:
BACKGROUND:

A solid foundation of epidemiologic, clinical and laboratory evidence underlies the current dietary recommendations for population-based prevention of coronary heart disease. Average blood cholesterol levels will decline with the consumption of less saturated fat and cholesterol than has been traditional in the United States. It is not clear, however, whether reductions in total fat intake are necessary as well. More research also is needed to define how best to provide a national food supply whose composition will enhance efforts to reduce coronary heart disease risk. Fatty acid investigations are especially critical, because this is an area in which the food industry has greater latitude in reformulating products according to current scientific evidence, dietary recommendations, and customer demand. Stearic acid, for example, may be suitable as a replacement for 'hard' fatty acids because it has relatively little effect on total blood cholesterol levels, but it may be rendered less suitable for this purpose if it accelerates the tendency of blood to clot. Similarly, hydrogenated vegetable oils are used as substitutes for saturated animal fats, but they contain trans-fatty acids that may raise low-density lipoprotein levels as do saturated fatty acids. In general, the mechanisms by which diet influences the eventual development of atherosclerosis through alterations in lipid and lipoprotein levels and metabolism, and through other factors such as hemostasis, still are not fully understood.

Human clinical nutrition studies, when feasible, are among the best research approaches for addressing the links between diet and atherosclerosis. Moreover, because of their great relevance to everyday life, their findings are quickly publicized. Often, however, such studies do not yield consistent or reproducible results. The resulting transmission of mixed messages to the scientific and lay communities seriously undermines both the credibility of nutrition research and the public's confidence in the possibility of obtaining reliable and practical advice on how to modify diet. Oat bran, with its rise and fall in the scientific and popular press as well as in the marketplace, is a good example of this phenomenon.

The lack of consistency among designs of clinical nutrition studies seeking to answer the same scientific question (for example, the influence of dietary fiber on serum cholesterol levels) means that their results cannot be readily compared. Some study designs are flawed, lacking adequate hypotheses and control groups. In addition, compliance in dietary studies is frequently less than ideal. Studies that allow participants to select and prepare their own food, even when adhering to an 'experimental' diet, frequently do not provide reliable results. Only in tightly controlled clinical settings, in which the participants receive all food from the experimental kitchen and are known to consume it, can the influence of poor compliance be minimized.

A further complication is that the actual composition of study diets may not be as intended due to natural variations in food sources and the vagaries of food composition databases. Such discrepancies can be sufficient to alter the results of the study and lead to false conclusions, yet research budgets seldom allow for the high cost of food composition analyses.

The typical small size of clinical nutrition studies has far-reaching effects. Because these studies are expensive and require great commitments of labor and space, it generally is very difficult for a single investigator funded by a traditional research grant to enroll, feed, and study more than 20 to 25 participants at one time. This imposes constraints on duration, design, and statistical power; consequently, many human nutrition studies lack sufficient power to detect biologically meaningful differences between groups or treatments. To avoid outside sources of variability that would further reduce study power, investigators usually make efforts to assemble a 'homogeneous' study population and minimize the number of factors that might impinge on the experimental design; thus, studies are most often conducted in young Caucasian males with average or even low plasma cholesterol levels. Not much is known, therefore, about how response to diet is affected by sex, age, race, co-morbid conditions (such as obesity), lipoprotein phenotype and other factors that would make the results more generalizable to the population at large. Furthermore, the mechanisms underlying the so-called 'hypo-responder' phenomenon, wherein individuals are presumed to be insensitive to the effects of diet on plasma lipid levels, cannot be elucidated unless individuals with a wide range of response are studied in adequate numbers.

The Arteriosclerosis, Hypertension, and Lipid Metabolism Advisory Committee recommended the development of the initiative at their February 1991 meeting. The National Heart, Lung, and Blood Advisory Council approved the concept at its September 1991 meeting.

DESIGN NARRATIVE:

The first protocol, conducted in 1993-1994, compared the effects of three diets varying in total fat (37 percent, 30 percent, and 26 percent) and saturated fat (16 percent, 9 percent, and 5 percent) on plasma lipoprotein and thrombogenic activity in 103 normal adults. Subjects consumed the three diets for eight weeks each. Ten meals per week were consumed on-site and all other food was packed for take-home use.

The second protocol, conducted in 1994-1995, examined lipoprotein levels and hemostatic parameters in 86 subjects having low high density lipoprotein levels and/or high triglyceride levels and/or high insulin levels and consuming for seven weeks each one of three diets: a typical American diet, a high monounsaturated fat diet, or a high carbohydrate diet.

DELTA also expended considerable effort in the field of food composition analysis. Menus were analyzed chemically to verify their composition and to ensure that the nutrient content did not differ significantly among field centers and diet periods. Food composition analysis research was conducted at Virginia Polytechnic and State University in consortium with the University of North Carolina.

The study was active through August 31, 1999 under grant U01-HL-49644.

ELIGIBILITY:
Men and women with low HDL and/or high triglyceride levels and/or high insulin levels.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 1992-09; Primary Completion 1995-05 (Actual); Study Completion 1995-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Elmer — University of Minnesota; Penny Kris-Etherton — Penn State University; Paul Roheim — Louisiana State University Medical Center; Henry Ginsberg — Columbia University

REFERENCES:
- [Background] Ginsberg HN. New directions in dietary studies and heart disease: the National Heart, Lung and Blood Institute sponsored Multicenter Study of Diet Effects on Lipoproteins and Thrombogenic Activity. Adv Exp Med Biol. 1995;369:241-7. doi: 10.1007/978-1-4615-1957-7_23. PMID 7598013
- [Background] Dennis BH, Stewart P, Wang CH, Champagne C, Windhauser M, Ershow A, Karmally W, Phillips K, Stewart K, Van Heel N, Farhat-Wood A, Kris-Etherton PM. Diet design for a multicenter controlled feeding trial: the DELTA program. Delta Research Group. J Am Diet Assoc. 1998 Jul;98(7):766-76. doi: 10.1016/s0002-8223(98)00173-4. PMID 9664917
- [Background] Lefevre M, Ginsberg HN, Kris-Etherton PM, Elmer PJ, Stewart PW, Ershow A, Pearson TA, Roheim PS, Ramakrishnan R, Derr J, Gordon DJ, Reed R. ApoE genotype does not predict lipid response to changes in dietary saturated fatty acids in a heterogeneous normolipidemic population. The DELTA Research Group. Dietary Effects on Lipoproteins and Thrombogenic Activity. Arterioscler Thromb Vasc Biol. 1997 Nov;17(11):2914-23. doi: 10.1161/01.atv.17.11.2914. PMID 9409276
- [Background] Reed RG, Kris-Etherton P, Stewart PW, Pearson TA. Variation of lipids and lipoproteins in premenopausal women compared with men and postmenopausal women. DELTA (Dietary Effects on Lipoproteins and Thrombogenic Activity) Investigators. Metabolism. 2000 Sep;49(9):1101-5. doi: 10.1053/meta.2000.8603. PMID 11016887
- [Background] Ginsberg HN, Kris-Etherton P, Dennis B, Elmer PJ, Ershow A, Lefevre M, Pearson T, Roheim P, Ramakrishnan R, Reed R, Stewart K, Stewart P, Phillips K, Anderson N. Effects of reducing dietary saturated fatty acids on plasma lipids and lipoproteins in healthy subjects: the DELTA Study, protocol 1. Arterioscler Thromb Vasc Biol. 1998 Mar;18(3):441-9. doi: 10.1161/01.atv.18.3.441. PMID 9514413
- [Background] Phillips KM, Tarrago-Trani MT, Grove TM, Grun I, Lugogo R, Harris RF, Stewart KK. Simplified gravimetric determination of total fat in food composites after chloroform-methanol extraction. Journal of American Oil Chemists' Society 74(2): 137-142, 1997.
- [Background] Mustad VA, Etherton TD, Cooper AD, Mastro AM, Pearson TA, Jonnalagadda SS, Kris-Etherton PM. Reducing saturated fat intake is associated with increased levels of LDL receptors on mononuclear cells in healthy men and women. J Lipid Res. 1997 Mar;38(3):459-68. PMID 9101427
- [Background] Phillips KM, Tarrago-Trani MT, Stewart KK. Phytosterol content of experimental diets differing in fatty acid composition. Food Chemistry 64(3): 415-422, 1999. https://www.sciencedirect.com/science/article/pii/S0308814698000909
- [Background] Berglund L, Oliver EH, Fontanez N, Holleran S, Matthews K, Roheim PS, Ginsberg HN, Ramakrishnan R, Lefevre M. HDL-subpopulation patterns in response to reductions in dietary total and saturated fat intakes in healthy subjects. Am J Clin Nutr. 1999 Dec;70(6):992-1000. doi: 10.1093/ajcn/70.6.992. PMID 10584043
- [Background] Kris-Etherton PM, Pearson TA, Wan Y, Hargrove RL, Moriarty K, Fishell V, Etherton TD. High-monounsaturated fatty acid diets lower both plasma cholesterol and triacylglycerol concentrations. Am J Clin Nutr. 1999 Dec;70(6):1009-15. doi: 10.1093/ajcn/70.6.1009. PMID 10584045
- [Background] Aussel C, Fehlmann M. Effect of alpha-fetoprotein on arachidonic acid metabolism in a human T-cell line. Immunol Lett. 1987 Jan;14(2):133-7. doi: 10.1016/0165-2478(87)90092-7. PMID 2438210
- [Derived] Kris-Etherton PM, Stewart PW, Ginsberg HN, Tracy RP, Lefevre M, Elmer PJ, Berglund L, Ershow AG, Pearson TA, Ramakrishnan R, Holleran SF, Dennis BH, Champagne CM, Karmally W; DELTA Investigators. The Type and Amount of Dietary Fat Affect Plasma Factor VIIc, Fibrinogen, and PAI-1 in Healthy Individuals and Individuals at High Cardiovascular Disease Risk: 2 Randomized Controlled Trials. J Nutr. 2020 Aug 1;150(8):2089-2100. doi: 10.1093/jn/nxaa137. PMID 32492148